CLINICAL TRIAL: NCT00658125
Title: Modulation of Cognitive Function Using Electrical Brain Stimulation in Patients With Early Alzheimer Disease
Brief Title: Deep Brain Stimulation (DBS) for Alzheimer's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Andres M. Lozano, Professor of Surgery, University Health Network, Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-0095-B
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Experimental (Experimental)
  Interventions: Procedure: Bilateral fornix DBS implantation,

INTERVENTIONS:
Procedure: Bilateral fornix DBS implantation, — Fornix DBS for Alzheimer Disease
  Other Names: DBS

SUMMARY:
Background: Alzheimer disease (AD) is a debilitating brain disorder that affects over 4.75 million people in the US and Canada. People with AD have difficulty remembering general facts and previously experienced autobiographical events. Animal and human research demonstrates that this type of memory depends on neural function within specific brain areas, and that it may be possible to enhance memory with electrical stimulation of these brain areas. We have recently shown that deep brain stimulation (DBS) of a brain area called the fornix enhances memory in a human.

Hypotheses: We hypothesize that fornix DBS will safely enhance memory in early AD patients by activating memory circuits in the brain.

Methods: Six early AD patients will take part in a phase I clinical study over a 1-year period. The study involves bilateral fornix DBS implantation, detailed neuropsychological and neurological testing, and brain imaging to detect alterations in brain activity induced by stimulation. These assessments will occur one month before surgery, then again at one month, 6 months, and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 to 80 years old, who
* Satisfy the diagnostic criteria for probable AD,
* Have received the diagnosis of AD within the past 2 years,
* Have a CDR of 0.5 or 1.0, and
* Score between 20 and 28 on the Mini Mental State Examination

Exclusion Criteria:

* Pre-existing structural brain abnormalities,
* Other neurologic or psychiatric diagnoses, or
* Medical comorbidities that would preclude them from undergoing surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2010-06-30 (Actual); Study Completion 2010-06-30 (Actual)

PRIMARY OUTCOMES:
memory performance on neuropsychological tests | one year

CONTACTS AND LOCATIONS:
Overall Officials: Adrian W Laxton, MD, Study Director — Toronto Western Research Institute; Andres M Lozano, MD, PhD, Principal Investigator — Toronto Western Research Institute; David Tang-Wai, MD, Principal Investigator — Toronto Western Research Institute
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hamani C, McAndrews MP, Cohn M, Oh M, Zumsteg D, Shapiro CM, Wennberg RA, Lozano AM. Memory enhancement induced by hypothalamic/fornix deep brain stimulation. Ann Neurol. 2008 Jan;63(1):119-23. doi: 10.1002/ana.21295. PMID 18232017